CLINICAL TRIAL: NCT03154255
Title: GOOD-DAY: Efficacy of Gamification of an educatiOnal Training tO meDiterranean Diet on Weight and Metabolic Control in pAediatric obesitY: a Pilot Open-label Randomized Controlled Trial
Brief Title: GOOD-DAY Trial in Paediatric Obesity
Acronym: GOOD-DAY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliero Universitaria Maggiore della Carita (Other)
Responsible Party: Principal Investigator, Flavia Prodam, Assoc. Professor in Clinical Nutrition, Azienda Ospedaliero Universitaria Maggiore della Carita
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CE 50/17
Record Dates: First submitted 2017-05-02; First posted 2017-05-16 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2021-08

CONDITIONS: Obesity, Childhood
Keywords: Obesity; Paediatric; Mediterranean diet; Gamification; Insulin-resistance
MeSH Terms: conditions — Pediatric Obesity; Obesity; Insulin Resistance

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mediterranean Style-Diet Group (Experimental): These subjects will receive a standard diet according to routine clinical practice + a 30 minutes Mediterranean-Style Diet educational training with explanation of Mediterranean pyramid + gamification to Mediterranean diet inside the Hospital and at home throughout "The Mediterranean Goose".
  Interventions: Behavioral: Mediterranean-Style Diet Educational Training
- Standard Diet Group (No Intervention): These subjects will receive Standard Diet according to routine care and practice. The standard diet will be distributed with 55-60% of carbohydrates (45-50% complex and no more than 10% refined and processed sugars), 25-30% lipids and 15% proteins, and will be performedin accordance with the calories of an isocaloric balanced diet calculated throughout the Italian LARN Guidelines for age and gender (Società Italiana di Nutrizione Umana, 2014), inspired to Mediterranean pyramid.

INTERVENTIONS:
Behavioral: Mediterranean-Style Diet Educational Training — The intervention consists in a standard diet according to routine clinical practice + a 30 minutes Mediterranean-Style Diet educational training with explanation of Mediterranean pyramid + gamification to Mediterranean diet inside the Hospital and at home throughout "The Mediterranean Goose".
  Arms: Mediterranean Style-Diet Group

SUMMARY:
Alongside efforts in public health and policy to reverse the childhood obesity epidemic, medical providers seek to play effective roles in prevention and treatment. Limited interventional studies with effective long-term maintenance of weight loss in children are available. Moreover, interventions should focus on modifying lifestyle, by improving also ludic educational training. In fact, the knowledge, attitudes, behaviors and skills developed through effective health programs may result in a better quality of life and empower children to make correct choices to promote the health of the individual the family and the community. For this reason, in a cohort of obese pediatric subjects with visceral adiposity, the aim of the study is to assess the efficacy of an educational training inspired to Mediterranean diet and based on gamification (as "The Mediterranean Goose") with respect to a conventional treatment on weight loss and improvement of cardio-metabolic risk factors.

DETAILED DESCRIPTION:
Study design: A single-center pilot open-label randomized control trial. Population: The study will comprise a total of 60 subjects of both sexes, between 10 and 18 years of age, obese, according to the IOTF criteria (Cole TJ et al., 2000) and with visceral adiposity, as waist circumference ≥ 90th percentile (Cook S et al., 2003 - Cruz ML, Goran MI, 2004 - de Ferranti SD et al., 2004), diet naïve or with failure of weight loss (defined as -1 kg/m2 BMI in 1 year).

Inclusion/ Exclusion criteria (see Eligibility Criteria). Intervention: Patients will be randomized in a open-label, into two groups homogeneous for number and sex of the subjects. One group (group SD) will receive Standard Diet according to routine care and practice, and one group (group SD+MSD) will receive a standard diet according to routine clinical practice + a 30 minutes Mediterranean-Style Diet educational training with explanation of Mediterranean pyramid + gamification to Mediterranean diet inside the Hospital and at home throughout "The Mediterranean Goose".

Dietary restriction: Thestandard diet will be distributed with 55-60% of carbohydrates (45-50% complex and no more than 10% refined and processed sugars), 25-30% lipids and 15% proteins, and will be performedin accordance with the calories of an isocaloric balanced diet calculated throughout the Italian LARN Guidelines for age and gender (Società Italiana di Nutrizione Umana, 2014), inspired to Mediterranean pyramid.The standard diet will be given as diet plans in writing, after explanation by a well-trained and experienced clinical paediatric endocrinologist.

Education in Hospital: As well as receiving the aforementioned recommendations, the SD+MSD group will also receive a simple visual guide of Mediterranean food pyramid explained by a dietitian/nutritionist for 30 minutes (Bach-Faig A et al., 2011).

Gamification: The MSD Group will be involved inside the Hospital in an educational and playful training playing to "The Mediterranean Goose" in the ludic area of the Pediatric Department; this game has been proposed in an educational project known as "Mediterranean diet and enhancement of traditional foodstuff - MedDiet", founded by European Union in the framework of the ENPI CBC Mediterranean Sea Basin Programme (www.med-diet.eu). This material will be given to the family for continue to play also at home.

Physical activity: all subjects will receive general recommendations about performing physical activity. Exercise will be conducted daily and will consist of 30 minutes of aerobic physical activity.

Randomization: Alternately per week, participants will be randomly assigned in a 1:1 to one of the two dietary intervention groups.

Timing: Patients will be evaluated firstly at time of enrollment (V0) and, during the first 2 weeks of study (V1), biochemical and ultrasound evaluations will be completed. During the year of intervention, patients will be evaluated after 3 months, 6 months and 12 months (V2, V3, V4).The following anthropometric measures, biochemical and ultrasound evaluations and questionnaires will be obtained:

1. Anthropometric measures:

   * height (V0, V2, V3, V4);
   * weight (V0, V2, V3, V4);
   * body mass index (BMI; Kg/m2) (V0, V2, V3, V4);
   * waist and hip circumferences (V0, V2, V3, V4) for the calculation of the following ratios: waist/hip, waist/height;
   * Tanner stage (V0, V2, V3, V4) (Tanner JM, 1961);
   * blood pressure and heart rate (V0, V2, V3, V4).
2. Biochemical evaluations (after a 12-h overnight fast): CBC with formula, serum insulin-like growth factor 1 (IGF1, ng/mL), 25-hydroxy (OH) vitamin D (ng/mL), uric acid (mg/dL), alkaline phosphatase (U/L), ACTH (pg/mL), cortisol (microg/dL), TSH (uuI/mL), fT4 (ng/dL) (V1, V3, V4); aspartate aminotransferase (AST, IU/L), alanine aminotransferase (ALT, IU/L); AST-to-ALT ratio will be calculated as the ratio of AST (IU/L) and ALT(IU/L)(V1, V3, V4); serum creatinine concentration (mg/dL) will be measured with the enzymatic method; according to the NKF-K/DOQI Guidelines for CKD in children and adolescents (Hogg RJ et al., 2003), the eGFR will be calculated using updated Schwartz's formula (Schwartz GJ et al., 2009): eGFR (mL/min/1.73 m2) = [0.413 x patient's height (cm)] / serum creatinine (mg/dL)(V1, V3, V4); glucose (mg/dL), insulin (μUI/mL); insulin-resistance (IR) will be calculated using the formula of Homeostasis Model Assessment (HOMA)-IR: (insulin [mU/L] x glucose [mmol/lL) / 22.5)(V1, V3, V4); lipid profile: total cholesterol (mg/dL), High-Density Lipoprotein (HDL)-cholesterol (mg/dL), triglycerides (mg/dL); Low-Density Lipoprotein (LDL)-cholesterol will be calculated by the Friedwald formula and non-HDL (nHDL)-cholesterol will be also calculated(V1, V3, V4); oral glucose tolerance test (OGTT: 1.75 g of glucose solution per kg, maximum 75 g) and samples willbe collected for the determination of glucose and insulin every 30 min. The area under the curve (AUC) for parameters after OGTT will be calculated according to the trapezoidal rule. Insulin sensitivity at fasting and during OGTT will be calculated as the formula of the Quantitative Insulin-Sensitivity Check Index (QUICKI) and Matsuda index (ISI). The stimulus for insulin secretion in the increment in plasma glucose as insulinogenic index will be calculated as the ratio of the changes in insulin and glucose concentration from 0 to 30 min (InsI). Βeta-cell compensatory capacity will be evaluated by the disposition index defined as the product of the ISI and InsI (DI) (Kahn SE et al., 1993)(V1, V4); a collection at rest of first-morning urine sample. Physical and chemical urinalysis; urine albumin (mg/L) will be determined by an advanced immunoturbidimetric assay and urine creatinine (mg/dL) will be measured using the enzymatic method. Urine albumin to creatinine ratio (u-ACR - mg/g), will be calculated using the following formula: [urine albumin (mg/dL) / urine creatinine (mg/dL)] x 1000. For these calculations both albumin and creatinine will be in the same unit. The subjects whose urine will be found positive, they will undergo a collection of two more samples and will be considered the u-ACR mean value of these (V1, V3, V4).
3. Ultrasound evaluations:

   * liver ultrasound(V1, V4);
   * echocardiography and carotid sonography(V1, V4).
4. Nutritional and physical activity measurements:

   * KIDMED questionnaire for children and adolescents; the index comprises 16 yes or no questions (Serra-Majem L et al., 2004), and the total score of the KIDMED index ranged from -4 to 12 and is classified into 3 levels: 1)≥8: optimal Mediterranean diet; 2) 4-7: improvement is needed to adjust intake to the Mediterranean diet; 3) ≤3: very low diet quality; the Italian version is reported and approved by Istituto Superiore Sanità in Rapporti ISTISAN 12/42(Istituto Superiore della Sanità, Rapporti ISTISAN 12/42, 2012)(V0, V2, V3, V4);
   * the Food Frequency Questionnaire section of the Children's Eating Habits Questionnaire (CEHQ-FFQ), performed by Identification and prevention of Dietary and lifestyle-induced health Effects In Children and infantS (IDEFICS) study, on which parents or other caregivers will be asked to report the number of meals the children usually consumed at home or at other people's homes, such as of grandparents and friends, in a typical week of the previous month (Huybrechts I et al., 2011) (V0, V2, V3, V4);
   * 24-hour recall and a list of all foods and constituents included in the Dietary Inflammatory Index (DII) along with the respective adjusted score will be evaluated. Food- and constituent-specific scores will be multiplied by the intake for each subject. and then will be summed to create the overall Inflammatory Index score (Cavicchia PP et al., 2009 - Shivappa N et al., 2014) (V0, V2, V3, V4);
   * the Mediterranean Adequacy Index (MAI) will be obtained by dividing the sum of the percentage of total energy from typical Mediterranean food groups by the sum of the percentage of total energy from non-typical Mediterranean food groups, according to the following equation (Alberti-Fidanza A, Fidanza F, 2004) (V0, V2, V3, V4);
   * the International Physical Activity Questionnaire (IPAQ) developed, validated for Italian adolescents (IPAQ-A) will be developed; It covers four domains of physical activity: (1) school-related physical activity, including activity during physical education classes and breaks, (2) transportation, (3) housework and (4) leisure time (Hagstromer M et al., 2008 - Mannocci A et al, Accepted to Minerva Pediatrica) (V0, V2, V3, V4).

Outcomes (see Outcome Measures). Information retrieval: A case report form (CRF) will be completed for each subject included in the study. The source documents will be the hospital's or the physician's chart.

Statistical e sample size: A sample of 60 individuals (30 in each group) has been estimated to be sufficient to demonstrate a difference of 0.4kg/m2 in BMISDS with a SD of 0.65 (Prodam F et al, 2013) with 90% power and a significance level of 95% and a drop-out rate of 20% using the Student test. Statistical significance will be assumed at P< 0.05. The statistical analysis will be performed with SPSS for Windows version 17.0 (SPSS Inc., Chicago, IL, USA).

Organization characteristics: The study will be conducted at the Pediatric Endocrine Service of Division of Pediatrics, Department of Health Sciences, University of Piemonte Orientale, in Novara.

All blood samples will be measured evaluated using standardized methods in the Hospital's Chemistry Laboratory, previously described (Prodam F et al., 2014 - Prodam F et al., 2016).

Good Clinical Practice: The protocol will be conducted in accordance with the declaration of Helsinki. Informed consent will be obtained from all parents prior to the evaluations after careful explanations to each patient.

ELIGIBILITY:
Inclusion Criteria:

* obesity, according to the IOTF criteria;
* waist circumference ≥ 90th percentile;
* diet naïve or with failure of weight loss (defined as -1 kg/m2 BMI in 1 year).

Exclusion Criteria:

* specific causes of endocrine or genetic obesity;
* type 1 diabetes;
* previous kidney diseases.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2017-10-03 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Change in weight - weight loss | Change from Baseline BMI at 3 months, 6 months and 12 months
  Variation of body mass index (BMI)

SECONDARY OUTCOMES:
Metabolic control | Change from Baseline HOMA-IR at 3 months, 6 months and 12 months
  Improvement of cardio-metabolic risk factors: insulin resistance (HOMA-IR)
Metabolic control | Change from Baseline lipid profile at 3 months, 6 months and 12 months
  Improvement of cardio-metabolic risk factors: lipid profile
Metabolic control | Change from Baseline blood pressure at 3 months, 6 months and 12 months
  Improvement of cardio-metabolic risk factors: arterial hypertension
Adherence to Mediterranean Diet | Change from Baseline KIDMED Index at 3 months, 6 months and 12 months
  Adherence to Mediterranean Diet, evaluating food and habits questionnaires

CONTACTS AND LOCATIONS:
Locations (1):
- Pediatric Endocrine Service of AOU Maggiore della Carità of Novara; SCDU of Pediatrics, Department of Health Sciences, University of Eastern Piedmont, Novara, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cole TJ, Lobstein T. Extended international (IOTF) body mass index cut-offs for thinness, overweight and obesity. Pediatr Obes. 2012 Aug;7(4):284-94. doi: 10.1111/j.2047-6310.2012.00064.x. Epub 2012 Jun 19. PMID 22715120
- [Background] Cook S, Weitzman M, Auinger P, Nguyen M, Dietz WH. Prevalence of a metabolic syndrome phenotype in adolescents: findings from the third National Health and Nutrition Examination Survey, 1988-1994. Arch Pediatr Adolesc Med. 2003 Aug;157(8):821-7. doi: 10.1001/archpedi.157.8.821. PMID 12912790
- [Background] Cruz ML, Goran MI. The metabolic syndrome in children and adolescents. Curr Diab Rep. 2004 Feb;4(1):53-62. doi: 10.1007/s11892-004-0012-x. PMID 14764281
- [Background] de Ferranti SD, Gauvreau K, Ludwig DS, Neufeld EJ, Newburger JW, Rifai N. Prevalence of the metabolic syndrome in American adolescents: findings from the Third National Health and Nutrition Examination Survey. Circulation. 2004 Oct 19;110(16):2494-7. doi: 10.1161/01.CIR.0000145117.40114.C7. Epub 2004 Oct 11. PMID 15477412
- [Background] Società Italiana di Nutrizione Umana.(2014).Livelli di assunzione raccomandati di energia e nutrienti per la popolazione italiana (LARN). Milan, Italy: S.I.N.U.
- [Background] Bach-Faig A, Berry EM, Lairon D, Reguant J, Trichopoulou A, Dernini S, Medina FX, Battino M, Belahsen R, Miranda G, Serra-Majem L; Mediterranean Diet Foundation Expert Group. Mediterranean diet pyramid today. Science and cultural updates. Public Health Nutr. 2011 Dec;14(12A):2274-84. doi: 10.1017/S1368980011002515. PMID 22166184
- [Background] Tanner JM. (1961). Growth at adolescence. 2 edn. Oxford: Blackwell Scientific Publications
- [Background] Hogg RJ, Furth S, Lemley KV, Portman R, Schwartz GJ, Coresh J, Balk E, Lau J, Levin A, Kausz AT, Eknoyan G, Levey AS; National Kidney Foundation's Kidney Disease Outcomes Quality Initiative. National Kidney Foundation's Kidney Disease Outcomes Quality Initiative clinical practice guidelines for chronic kidney disease in children and adolescents: evaluation, classification, and stratification. Pediatrics. 2003 Jun;111(6 Pt 1):1416-21. doi: 10.1542/peds.111.6.1416. PMID 12777562
- [Background] Schwartz GJ, Munoz A, Schneider MF, Mak RH, Kaskel F, Warady BA, Furth SL. New equations to estimate GFR in children with CKD. J Am Soc Nephrol. 2009 Mar;20(3):629-37. doi: 10.1681/ASN.2008030287. Epub 2009 Jan 21. PMID 19158356
- [Background] Kahn SE, Prigeon RL, McCulloch DK, Boyko EJ, Bergman RN, Schwartz MW, Neifing JL, Ward WK, Beard JC, Palmer JP, et al. Quantification of the relationship between insulin sensitivity and beta-cell function in human subjects. Evidence for a hyperbolic function. Diabetes. 1993 Nov;42(11):1663-72. doi: 10.2337/diab.42.11.1663. PMID 8405710
- [Background] Serra-Majem L, Ribas L, Ngo J, Ortega RM, Garcia A, Perez-Rodrigo C, Aranceta J. Food, youth and the Mediterranean diet in Spain. Development of KIDMED, Mediterranean Diet Quality Index in children and adolescents. Public Health Nutr. 2004 Oct;7(7):931-5. doi: 10.1079/phn2004556. PMID 15482620
- [Background] Istituto Superiore della Sanità, Censi L, D'Addesa D, Galeone D et al. (2012). Studio ZOOM8: l'alimentazione e l'attività fisica dei bambini della scuola primaria. Rapporti ISTISAN 12/42.
- [Background] Huybrechts I, Bornhorst C, Pala V, Moreno LA, Barba G, Lissner L, Fraterman A, Veidebaum T, Hebestreit A, Sieri S, Ottevaere C, Tornaritis M, Molnar D, Ahrens W, De Henauw S; IDEFICS Consortium. Evaluation of the Children's Eating Habits Questionnaire used in the IDEFICS study by relating urinary calcium and potassium to milk consumption frequencies among European children. Int J Obes (Lond). 2011 Apr;35 Suppl 1:S69-78. doi: 10.1038/ijo.2011.37. PMID 21483425
- [Background] Cavicchia PP, Steck SE, Hurley TG, Hussey JR, Ma Y, Ockene IS, Hebert JR. A new dietary inflammatory index predicts interval changes in serum high-sensitivity C-reactive protein. J Nutr. 2009 Dec;139(12):2365-72. doi: 10.3945/jn.109.114025. Epub 2009 Oct 28. PMID 19864399
- [Background] Shivappa N, Steck SE, Hurley TG, Hussey JR, Hebert JR. Designing and developing a literature-derived, population-based dietary inflammatory index. Public Health Nutr. 2014 Aug;17(8):1689-96. doi: 10.1017/S1368980013002115. Epub 2013 Aug 14. PMID 23941862
- [Background] Alberti-Fidanza A, Fidanza F. Mediterranean Adequacy Index of Italian diets. Public Health Nutr. 2004 Oct;7(7):937-41. doi: 10.1079/phn2004557. PMID 15482621
- [Background] Hagstromer M, Bergman P, De Bourdeaudhuij I, Ortega FB, Ruiz JR, Manios Y, Rey-Lopez JP, Phillipp K, von Berlepsch J, Sjostrom M; HELENA Study Group. Concurrent validity of a modified version of the International Physical Activity Questionnaire (IPAQ-A) in European adolescents: The HELENA Study. Int J Obes (Lond). 2008 Nov;32 Suppl 5:S42-8. doi: 10.1038/ijo.2008.182. PMID 19011653
- [Background] Mannocci A, Masala D, Mei D, Tribuzio AM, Villari P, LA Torre G. International Physical Activity Questionnaire for Adolescents (IPAQ A): reliability of an Italian version. Minerva Pediatr (Torino). 2021 Oct;73(5):383-390. doi: 10.23736/S2724-5276.16.04727-7. Epub 2018 Jan 29. PMID 29381006
- [Background] Prodam F, Ricotti R, Agarla V, Parlamento S, Genoni G, Balossini C, Walker GE, Aimaretti G, Bona G, Bellone S. High-end normal adrenocorticotropic hormone and cortisol levels are associated with specific cardiovascular risk factors in pediatric obesity: a cross-sectional study. BMC Med. 2013 Feb 20;11:44. doi: 10.1186/1741-7015-11-44. PMID 23425018
- [Background] Prodam F, Savastio S, Genoni G, Babu D, Giordano M, Ricotti R, Aimaretti G, Bona G, Bellone S. Effects of growth hormone (GH) therapy withdrawal on glucose metabolism in not confirmed GH deficient adolescents at final height. PLoS One. 2014 Jan 30;9(1):e87157. doi: 10.1371/journal.pone.0087157. eCollection 2014. PMID 24498035
- [Background] Prodam F, Zanetta S, Ricotti R, Marolda A, Giglione E, Monzani A, Walker GE, Rampone S, Castagno M, Bellone S, Petri A, Aimaretti G, Bona G. Influence of Ultraviolet Radiation on the Association between 25-Hydroxy Vitamin D Levels and Cardiovascular Risk Factors in Obesity. J Pediatr. 2016 Apr;171:83-9.e1. doi: 10.1016/j.jpeds.2015.12.032. Epub 2016 Jan 12. PMID 26794470
- See also: "Mediterranean diet and enhancement of traditional foodstuff - MedDiet" — http://www.med-diet.eu